CLINICAL TRIAL: NCT00160108
Title: A Dietary Intervention- Randomized Controlled Trial (DIRECT) Study; BGU-Harvard-Robarts Collaboration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The S. Daniel Abraham International Center for Health and Nutrition (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other); University of Western Ontario, Canada (Other); Soroka University Medical Center (Other); Brigham and Women's Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); The Nuclear Research Center, Dimona (Unknown); Ben-Gurion University of the Negev (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DR300-3
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2006-09

CONDITIONS: Obesity; CHD
MeSH Terms: conditions — Obesity | interventions — Diet Therapy

INTERVENTIONS:
Behavioral: dietary intervention

SUMMARY:
Aim-to conduct a randomized clinical intervention study to compare three diets (low-fat, low-carbohydrate and Mediterranean diet) for weight loss

DETAILED DESCRIPTION:
Aim-to conduct a randomized clinical intervention study to compare three diets (low-fat, low-carbohydrate and Mediterranean diet) for weight loss

ELIGIBILITY:
Inclusion Criteria:

* BMI>27
* age>40
* History of CHD or diabetes in any age or BMI level

Exclusion Criteria:

* Pregnant or lactating women.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Serum creatinine > 3 mg/dl.
* Liver dysfunction ( ³ 2 fold level of ALT and AST enzymes).
* Participation in another trial in which active intervention is being received.
* Any intestinal problem that would prevent the patient from eating one of the test diets (for example, gastric stapling that might prevent consumption of vegetables).

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
weight loss

SECONDARY OUTCOMES:
CVD mediators measurements

CONTACTS AND LOCATIONS:
Overall Officials: Iris Shai, RD, PhD, Principal Investigator — Ben-Gurion University of the Negev; Meir J Stampfer, MD, DrPH, Study Chair — Departments of Epidemiology and Nutrition, Harvard School of Public Health, Boston, Massachusetts, USA; David Spence, MD, Study Chair — Stroke Prevention & Atherosclerosis Research Centre, Robarts Research Institute, London, Canada
Locations (1):
- Medical Center, The Nuclear Research Center, Dimona, Israel

REFERENCES:
- [Background] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Derived] Yaskolka Meir A, Tsaban G, Rinott E, Zelicha H, Schwarzfuchs D, Gepner Y, Rudich A, Shelef I, Bluher M, Stumvoll M, Ceglarek U, Isermann B, Kloting N, Keller M, Kovacs P, Qi L, Wang DD, Liang L, Hu FB, Stampfer MJ, Shai I. Individual response to lifestyle interventions: a pooled analysis of three long-term weight loss trials. Eur J Prev Cardiol. 2025 Nov 11;32(16):1660-1670. doi: 10.1093/eurjpc/zwaf308. PMID 40472282
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Derived] Yokose C, McCormick N, Rai SK, Lu N, Curhan G, Schwarzfuchs D, Shai I, Choi HK. Effects of Low-Fat, Mediterranean, or Low-Carbohydrate Weight Loss Diets on Serum Urate and Cardiometabolic Risk Factors: A Secondary Analysis of the Dietary Intervention Randomized Controlled Trial (DIRECT). Diabetes Care. 2020 Nov;43(11):2812-2820. doi: 10.2337/dc20-1002. Epub 2020 Sep 2. PMID 33082244
- [Derived] Zheng Y, Ceglarek U, Huang T, Li L, Rood J, Ryan DH, Bray GA, Sacks FM, Schwarzfuchs D, Thiery J, Shai I, Qi L. Weight-loss diets and 2-y changes in circulating amino acids in 2 randomized intervention trials. Am J Clin Nutr. 2016 Feb;103(2):505-11. doi: 10.3945/ajcn.115.117689. Epub 2016 Jan 20. PMID 26791187
- [Derived] Tirosh A, Golan R, Harman-Boehm I, Henkin Y, Schwarzfuchs D, Rudich A, Kovsan J, Fiedler GM, Bluher M, Stumvoll M, Thiery J, Stampfer MJ, Shai I. Renal function following three distinct weight loss dietary strategies during 2 years of a randomized controlled trial. Diabetes Care. 2013 Aug;36(8):2225-32. doi: 10.2337/dc12-1846. Epub 2013 May 20. PMID 23690533
- [Derived] Canfi A, Gepner Y, Schwarzfuchs D, Golan R, Shahar DR, Fraser D, Witkow S, Greenberg I, Sarusi B, Vardi H, Friger M, Stampfer MJ, Shai I. Effect of changes in the intake of weight of specific food groups on successful body weight loss during a multi-dietary strategy intervention trial. J Am Coll Nutr. 2011 Dec;30(6):491-501. doi: 10.1080/07315724.2011.10719995. PMID 22331684
- [Derived] Bluher M, Rudich A, Kloting N, Golan R, Henkin Y, Rubin E, Schwarzfuchs D, Gepner Y, Stampfer MJ, Fiedler M, Thiery J, Stumvoll M, Shai I. Two patterns of adipokine and other biomarker dynamics in a long-term weight loss intervention. Diabetes Care. 2012 Feb;35(2):342-9. doi: 10.2337/dc11-1267. Epub 2011 Dec 21. PMID 22190676
- [Derived] Leichtle AB, Helmschrodt C, Ceglarek U, Shai I, Henkin Y, Schwarzfuchs D, Golan R, Gepner Y, Stampfer MJ, Bluher M, Stumvoll M, Thiery J, Fiedler GM. Effects of a 2-y dietary weight-loss intervention on cholesterol metabolism in moderately obese men. Am J Clin Nutr. 2011 Nov;94(5):1189-95. doi: 10.3945/ajcn.111.018119. Epub 2011 Sep 21. PMID 21940598
- [Derived] Golan R, Tirosh A, Schwarzfuchs D, Harman-Boehm I, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Shai I; DIRECT Group. Dietary intervention induces flow of changes within biomarkers of lipids, inflammation, liver enzymes, and glycemic control. Nutrition. 2012 Feb;28(2):131-7. doi: 10.1016/j.nut.2011.04.001. Epub 2011 Aug 6. PMID 21820871
- [Derived] Shahar DR, Schwarzfuchs D, Fraser D, Vardi H, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ, Shai I; DIRECT Group. Dairy calcium intake, serum vitamin D, and successful weight loss. Am J Clin Nutr. 2010 Nov;92(5):1017-22. doi: 10.3945/ajcn.2010.29355. Epub 2010 Sep 1. PMID 20810979
- [Derived] Shai I, Spence JD, Schwarzfuchs D, Henkin Y, Parraga G, Rudich A, Fenster A, Mallett C, Liel-Cohen N, Tirosh A, Bolotin A, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; DIRECT Group. Dietary intervention to reverse carotid atherosclerosis. Circulation. 2010 Mar 16;121(10):1200-8. doi: 10.1161/CIRCULATIONAHA.109.879254. Epub 2010 Mar 1. PMID 20194883
- [Derived] Shai I, Schwarzfuchs D, Henkin Y, Shahar DR, Witkow S, Greenberg I, Golan R, Fraser D, Bolotin A, Vardi H, Tangi-Rozental O, Zuk-Ramot R, Sarusi B, Brickner D, Schwartz Z, Sheiner E, Marko R, Katorza E, Thiery J, Fiedler GM, Bluher M, Stumvoll M, Stampfer MJ; Dietary Intervention Randomized Controlled Trial (DIRECT) Group. Weight loss with a low-carbohydrate, Mediterranean, or low-fat diet. N Engl J Med. 2008 Jul 17;359(3):229-41. doi: 10.1056/NEJMoa0708681. PMID 18635428